CLINICAL TRIAL: NCT00388518
Title: A Randomized, Double-blind Study to Investigate the Effect of Aleglitazar on Glycemic Control in Patients With Type 2 Diabetes Mellitus.
Brief Title: A Study of Aleglitazar in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM17864
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Actos (Active Comparator)
  Interventions: Drug: Actos
- Aleglitazar 1 (Experimental)
  Interventions: Drug: aleglitazar
- Aleglitazar 2 (Experimental)
  Interventions: Drug: aleglitazar
- Aleglitazar 3 (Experimental)
  Interventions: Drug: aleglitazar
- Aleglitazar 4 (Experimental)
  Interventions: Drug: aleglitazar
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Actos — 45mg po daily
  Arms: Actos
Drug: Placebo — po daily
  Arms: Placebo
Drug: aleglitazar — Administered po daily, at ascending doses with a starting dose (arm 1) of 0.05mg.
  Arms: Aleglitazar 1; Aleglitazar 2; Aleglitazar 3; Aleglitazar 4

SUMMARY:
This 6 arm study will assess the efficacy, safety, tolerability and pharmacokinetics of aleglitazar therapy in patients with Type 2 diabetes. Patients will be randomised to one of 6 treatment arms, to receive one of 4 doses of aleglitazar, Actos as an open-label active comparator, or placebo. Aleglitazar will be administered starting from a dose of 0.05mg po daily, and Actos will be administered at a dose of 45mg once daily. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes, diagnosed >=1 month of screening;
* either drug-naive, or pretreated with a maximum of 2 oral antihyperglycemic agents at submaximal doses;
* HbA1c <=10.0% at screening, and 7.0-10.0% at pre-randomisation visit.

Exclusion Criteria:

* type 1 diabetes;
* currently or previously treated with insulin, a thiazolidinedione, or a dual Peroxisome Proliferator Activated Receptor (PPAR) agonist;
* clinically significant cardiovascular disease;
* Congestive Heart Failure (CHF) New York Heart Association (NYHA) 3-4.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in Hemoglobin A1c (HbA1c) | 16 weeks

SECONDARY OUTCOMES:
Absolute change from baseline in Fasting Plasma Glucose (FPG), HbA1c response rate, insulin sensitivity, beta cell function and cardiovascular markers. | 16 weeks
Adverse Events (AEs), laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (47):
- United States (17):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Palm Springs, California
  - San Diego, California
  - Chiefland, Florida
  - Hollywood, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Olive Branch, Mississippi
  - Hamilton, New Jersey
  - New Hyde Park, New York
  - Johnson City, Tennessee
  - Spokane, Washington
- Greece (2):
  - Athens
  - Thessaloniki
- Hong Kong, Hong Kong
- Italy (9):
  - Bologna
  - Genova
  - Napoli
  - Olbia
  - Pavia
  - Perugia
  - Roma
  - Siena
  - Torino
- Mexico (8):
  - Aguascalientes
  - Chihuahua City
  - Cuernavaca
  - Durango
  - Guadalajara
  - Mexico City
  - Monterrey
  - Pachuca
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Galati
  - Ploieşti
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Saratov
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Niš

REFERENCES:
- [Derived] Henry RR, Lincoff AM, Mudaliar S, Rabbia M, Chognot C, Herz M. Effect of the dual peroxisome proliferator-activated receptor-alpha/gamma agonist aleglitazar on risk of cardiovascular disease in patients with type 2 diabetes (SYNCHRONY): a phase II, randomised, dose-ranging study. Lancet. 2009 Jul 11;374(9684):126-35. doi: 10.1016/S0140-6736(09)60870-9. Epub 2009 Jun 8. PMID 19515415